CLINICAL TRIAL: NCT01623635
Title: Intraperitoneal Atomization of Ropivacaine During Gynecologic Laparoscopic Surgery: Impact on Pain, Opioid Use and Length of Recovery Room Stay
Brief Title: Intraperitoneal Atomization of Ropivacaine During Gynecologic Laparoscopic Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-004203-20
Record Dates: First submitted 2012-02-15; First posted 2012-06-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Case - adnexal (Experimental)
  Interventions: Drug: Ropivacaine
- placebo - adnexal (Placebo Comparator)
  Interventions: Drug: placebo (normal saline)
- case - uterine (Experimental)
  Interventions: Drug: Ropivacaine
- placebo - uterine (Placebo Comparator)
  Interventions: Drug: placebo (normal saline)

INTERVENTIONS:
Drug: Ropivacaine — ADMINISTRATION OF STUDY DRUG All surgical port sites will be injected with 2 ml/each study drug prior to trocar insertion
  Immediately following insufflation the Optispray surgical spray device will be inserted into the abdomen and directed towards the diaphragms, dome of inflated abdomen, bowel peritoneum and surgical dissection site and the study drug will be delivered as an atomized spray in the following volumes:
  * each subdiaphragmatic area 3.5 ml + 3.5ml
  * surgical dissection site 3 ml
  * diffusely across the peritoneal surface (dome of the abdomen and surface of the visible bowel) 7 ml. At the end of the case the remaining medication with be atomized again onto the same areas, using the same volumes.
  At the end of the case - this process will be repeated with the remaining drug (no repeat port site injections).
  Arms: Case - adnexal; case - uterine
Drug: placebo (normal saline) — ADMINSTRATION OF PLACEBO All surgical port sites will be injected with 2 ml/each placebo prior to trocar insertion
  Immediately following insufflation the Optispray surgical spray device will be inserted into the abdomen and directed towards the diaphragms, dome of inflated abdomen, bowel peritoneum and surgical dissection site and the placebo will be delivered as an atomized spray in the following volumes:
  * each subdiaphragmatic area 3.5 ml + 3.5ml
  * surgical dissection site 3 ml
  * diffusely across the peritoneal surface (dome of the abdomen and surface of the visible bowel) 7 ml. At the end of the case the remaining placebo with be atomized again onto the same areas, using the same volumes.
  At the end of the case - this process will be repeated with the remaining placebo (no repeat port site injections).
  Arms: placebo - adnexal; placebo - uterine

SUMMARY:
Pain following laparoscopic surgery continues to be a clinically important problem with 80% or more patients requiring opioid analgesia post-operatively to control their pain. By reducing this surgical complication patients can experience less discomfort and be discharged from the recovery room more rapidly leading to reduced resource utilization and expense.

HYPOTHESIS: Post-operative pain after laparoscopic procedures could be treated by topical anesthetics sprayed directly into the abdomen (inside the abdominal cavity, on the nerve endings of the visceral peritoneal lining and diaphragm surface) via the surgical incision METHODS: Randomized controlled trial on use of topical anesthetic (namely 0.25% ropivacaine) delivered directly onto the target sites both at the beginning and the end of surgery in patients undergoing laparoscopic gynecologic procedure for uterine or adnexal benign pathology. The drug will be delivered using a CE approved delivery system that will direct a fine mist of drug directly to the areas of the peritoneal cavity that are theoretically the cause of post-op pain (diaphragms, peritoneal abdominal surface, surgical dissection site).

GOAL: to assess the efficacy of intraperitoneal topical anesthesia in reducing postoperative pain, opioid requirements in patients undergoing laparoscopic gynecologic procedure for uterine or adnexal benign pathology

DETAILED DESCRIPTION:
Introduction:

Laparoscopic surgery has replaced open surgical techniques for a large number of abdominal general surgical and gynecologic interventions. However pain following laparoscopic surgery continues to be a clinically important problem with 80% or more patients requiring opioid analgesia post-operatively to control their pain. Post-operative pain and to a lesser extent post-operative nausea and vomiting (PONV) are the main factors leading to delayed discharge from the surgical recovery room and from the hospital following most surgical cases. Hence, post-operative pain and PONV lead to increased costs of care. By reducing these surgical complications patients can be discharged from the recovery room more rapidly leading to reduced resource utilization and expense. This is especially true for routine surgical cases (laparoscopic cholecystectomy -gallbladder removal, gynecologic procedures, gastric surgery) that have the potential for same day surgery and discharge to home if their pain can be adequately treated. It also applies to inpatient cases where superior pain control and less PONV require less nursing care and potentially earlier discharge.

The origin of pain after laparoscopic surgery is multifactorial with pain arising from the incision site, direct trauma in the area of surgical dissection, peritoneal micro-tears and inflammation due stretching during insufflation and peritoneal and diaphragm irritation of from the residual CO2 remaining after the pneumoperitoneum is deflated. Because this pain is multifactorial - a multifactorial approach is needed. Although the somatic pain associated with the abdominal wall incision responds well to nerve blocks or opiate medications, visceral pain due to pneumoperitoneum induced stretching, compression, oxygen deprivation and inflammation during the surgery is less responsive to these interventions. However, visceral pain can be treated by topical anesthetics sprayed directly onto the nerve endings of the visceral peritoneal lining and diaphragm surface. This knowledge has resulted in extensive research studying the effects of applying topical anesthetics to the peritoneal surface during laparoscopic surgery in an effort to reduce post-operative pain and its attendant complications. Fairly clear conclusions can be drawn from review of the research investigating topical anesthetic application to the peritoneum, diaphragms and surgical site: they effectively reduce postoperative pain and opioid use. They do not have any of the adverse effects of systemically administered opioids such as sedation, respiratory depression, nausea, or GI dysmotility. They are safe and relatively inexpensive. Their use results in earlier progression to ambulation, less shoulder tip pain, less post-operative nausea and vomiting, earlier discharge from the recovery room and in some studies earlier discharge from the hospital.

Despite this research and international recommendations to use this therapy topical anesthetic application during laparoscopic surgery is not routinely used by most general or obstetrical surgeons. There are probably two inter-related reasons for this lack of adoption of this simple concept. First, no simple method exists for delivering topical anesthetics to the peritoneal surface. Most studies diluted the drug with large volumes of saline (making it less potent and less likely to work), then injected it into a trocar where gravity took the solution straight into the gravity dependent gutters. This type of delivery system would not be expected to optimize results of any topically active medication since the majority of the peritoneal surface is never exposed to the anesthetic. Secondly, the pain reductions reported in most topical anesthetic studies were positive but not impressive enough for surgeons to change practice. This marginal reduction in post-operative pain is probably due to these poor delivery systems with non-directed application of the drug and the great variations in drug concentrations, site of delivery, and timing of application. Studies that used more directed spray seem to show better results. A 2010 metaanalysis concludes that future studies should not be designed to determine if topical intraperitoneal local anesthesia is effective (this is already proven), rather this research should focus on optimization of the method of delivery (aerosolized), location of application, timing of drug delivery, and drug dose and concentration.

This study is designed to address these issues. The investigators will use topical anesthetic (namely 0.25% ropivacaine) delivered directly onto the target sites both at the beginning and the end of surgery. The drug will be delivered using an inexpensive delivery system that will direct a fine mist of drug directly to the areas of the peritoneal cavity that are theoretically the cause of post-op pain (diaphragms, peritoneal abdominal surface, surgical dissection site). Our primary goal is to assess the efficacy of intraperitoneal topical anesthesia in reducing postoperative pain, opioid requirements in patients undergoing laparoscopic gynecologic laparoscopic procedure for uterus or adnexal benign pathology.

Materials and Methods:

Design:

Prospective, randomized, double-blinded, placebo controlled trial stratified by pathology (uterus or adnexal benign).

Clinicaltrials.gov submission: This study design will be submitted to the clinicaltrials.gov prospective trials registry as required by many journals.

Patients:

Women scheduled for elective gynecologic laparoscopic procedure for uterus or adnexal benign pathology

Intervention:

Patients will be randomized to ropivicaine 0.25% 40 ml (100 mg) or placebo (NaCl 0.9%) according to a randomization list stratified by pathology delivered in the following fashion:

* the derma at the portal sites will each be injected with 2 ml of medication at the onset of the surgery (total volume 6 ml).
* following insufflation of the abdomen, half of the remaining ropivacaine will be atomized onto each subdiaphragmatic area (3.5ml + 3.5ml), onto the surgical dissection site (3 ml) and diffusely across the peritoneal surface (dome of the abdomen and surface of the visible bowel) (7ml). At the end of the case the remaining medication with be atomized again onto the same areas, using the same volumes.

Primary Outcome Measured:

1. Post-operative pain intensity (NRS score. NRS; 0 = no pain and 10 = worse pain possible) at 6h post-operatively.

Secondary Outcomes measured

1. Total post-operative opioid analgesic requirements in the first 48 hours post-operatively or until discharge
2. Post-operative rescue opioid analgesic requirements in the first 6h post-operatively
3. Post-operative pain intensity scores during the first 48 hours post-operatively or until discharge - measured at times 0, 1, 2, 4, 6, 10, 18, 24, 36, 48 hours
4. Post-operative shoulder pain (NRS score. NRS; 0 = no pain and 10 = worse pain possible) intensity scores during the first 48 hours post-operatively or until discharge - measured at times 0, 1, 2, 4, 6, 10, 18, 24, 36, 48 hours
5. Post-operative nausea and vomiting verbal description scores (0 = no symptoms, 1 = nausea, 2 = nausea and vomiting) - measured at times 0, 1, 2, 4, 6, 10, 18, 24, 36, 48 hours
6. Post-operative sedation scores (Sedation will be evaluated using a 6 point Ramsay sedation score: 1= anxious and agitated, 2 = cooperative, tranquil, oriented, 3 = responds only to verbal commands, 4 = asleep with brisk response to light stimulation, 5 = asleep without response to light stimulation, 6 = non-responsive) measured at times 0, 1, 2, 4, 6 hours
7. Time until discharge from recovery room
8. Time until discharge from hospital
9. Time until first flatus or bowel movement
10. Time until ambulation.

Study Drug:

Study drug: ropivacaine 0.25% (2,5 mg/ml - 100 mg total) a local anesthetic manufactured by Astra Zeneca (Basiglio, MI, Italy).

Placebo: Saline 0.9% (Fresenius Kabi, Isola della Scala, VR, Italy). Study Drug and Placebo will be provided free of charge by the manufacturing companies, which will not have any other role in the study.

Drug and placebo prepared under sterile conditions in a specific syringe in the O.R. by an O.R. nurse, which thereafter will not be involved in the surgical operation nor in the patient care in the recovery room.

Random sequence generation by a computer generated random number table will be used to randomize each vial. Records of placebo versus active drug will be kept by the O.R. coordinator, and not available to investigators until the end of study data analysis.

Study device:

Optispray surgical spray device [CE mark (0050)], manufactured by AbViser Medical, Salt Lake City, UT, U.S.A. will be provided free of charge by the manufacturing company, which will not have any other role in the study.

Procedure:

1. Potentially eligible patients will be screened and consented at the time of pre-operative surgical evaluation (the night prior or morning of surgery).

2. A standard anesthetic procedure will be conducted for all patients.

* Pre-medication with midazolam 0.03mg/kg I.V.
* Induction with propofol 2 mg/kg. Maintenance with propofol 6mg/kg/h I.V.
* Muscle relaxation with cisatracurium, reversal with neostigmine and atropine
* Intra-operative analgesia will be standardized and administered by the anesthesiologist to all patients:

  * Fentanyl 2mcg/kg I.V. at induction, then 2mcg/kg 5 min before surgical incision and 2mcg/kg 30 minutes prior to the end of surgery
  * Remifentanil 0.1-0.3 mcg/kg/min I.V.
  * Acetaminophen 1g I.V. and Ketoprofen 100 mg I.V. will be administered 30 minutes prior to the end of surgery 4. A standard intra-operative antiemetic (Ondansetron 4 mg I.V.) will be administered by anesthesia 15 minutes prior to end of surgery.

    5. All laparoscopies will be performed in a standardized fashion
    1. Pneumoperitoneum by open technique (insufflation pressure 20 mmHg)
    2. Insertion of 3 trocars
    3. Intraabdominal pressure maintained at 12 mmHg
    4. Uterine or ovarian surgical procedure in a standardized fashion

       6. All study drug delivery will be performed in a standardized fashion

    a. All port sites will be injected with 2 ml/each study drug prior to trocar insertion b. Immediately following insufflation the Optispray surgical spray device will be inserted into the abdomen and directed towards the diaphragms, dome of inflated abdomen, bowel peritoneum and surgical dissection site and the study drug will be delivered as an atomized spray in the following volumes:
* each subdiaphragmatic area 3.5 ml + 3.5ml
* surgical dissection site 3 ml
* diffusely across the peritoneal surface (dome of the abdomen and surface of the visible bowel) 7 ml. At the end of the case the remaining medication with be atomized again onto the same areas, using the same volumes.

  c. At the end of the case - this process will be repeated with the remaining drug (no repeat port site injections).

  7. Postoperative analgesics:
* patients will receive Acetaminophen 1g I.V. 6h after surgery, then acetaminophen 1g per os every 8h
* rescue analgesic will be Tramadol 100mg in 50 ml of 0.9% saline I.V., preceded by I.V. 0.01mg/kg droperidol.

  8. Rescue post-operative antiemetics:
* ondansetron 4mg I.V. (Maximal for 3 times/day)

Data Collection procedure Data will be collected by investigator and stored in the Dipartimento di Scienze Ginecologiche e della Riproduzione Umana. Electronic datasets will be prepared including only anonymous data. Statistical analysis will be performed using SPSS v.18 computer program (SPSS Inc., Chicago, IL, USA).

Risks to patient:

The only risk to the patient from this study is the risk of local anesthetic toxicity. The toxicity of local anesthetics includes seizures and ventricular arrhythmias. At the currently selected doses this is very low probability for the following reasons: the doses selected are below the toxic doses described by the package insert for injected ropivacaine, and yet this dose in not being injected rather it is being sprayed onto the peritoneal surface. While there is no question some of the drug will be absorbed, this will occur over time and the peak levels will not achieve that expected when a drug is injected I.V.. Finally, prior literature studies have used similar doses and do not describe any toxicity in their patients nor toxic serum concentrations when applied to the peritoneal surface.

Benefits to patient This procedure is already proven to reduce postoperative pain in numerous studies but is not routinely used. Therefore, the patient has a 50% probability of being delivered the active anesthetic drug and can reasonably expect to have less pain if they are in that arm of the study. Furthermore, if they have reduced pain and use fewer opiates they may have less nausea and they may be discharged from recovery room and possible from the hospital more rapidly.

Statistical Analysis The investigators will examine separately uterine surgical procedures and adnexal surgical procedures.

Sample size determination:

Pain reduction: The study intention is to show a CLINICALLY significant reduction in pain (not just statistically significant). This can be hard to define if they have relatively low baseline pain, but most patients with anything but very minor laparoscopic surgeries who have been studied in the past wake up with pain scores in the 4-6 range - 6 being more typical. A pain score reduction of 1.5 would be 25% or more pain reduction (and the investigators know from prior studies that 1.3 or 23% reduction is the lower limit of clinically significant pain reduction).

A sample size of 45 in each group (treatment vs control) will have 80% power to detect a difference in means of 1.500 (the difference between a Group 1 mean of 6.000 and a Group 2 mean of 4.500) assuming that the common standard deviation is 2.500 using a two group t-test with a 0.050 two-sided significance level.

Due to potential drop-outs, the investigators will include 50 patients in each group, for a total of 200 patients (100 undergoing uterine procedures and 100 undergoing adnexal procedures). Statistical analysis will be performed as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective laparoscopic surgical intervention for benign uterine or adnexal conditions

Exclusion Criteria:

* Less than 18 year old
* Pregnancy
* Prisoners
* Allergic/contraindications to topical anesthetics (Amides specifically)
* Allergic/contraindications to Opioids as a class
* Allergic/contraindications to acetaminophen
* Allergic/contraindications to Propofol
* Allergic/contraindications to NSAIDS
* Currently or within the last 30 days been prescribed an opiate medication
* History of drugs or alcohol abuse
* Chronic pain syndrome
* Suspected gynecologic malignancy
* Poor comprehension of written and spoken Italian for informed consent purpose

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain intensity | at 6h post-operatively
  NRS score. (NRS; 0 = no pain and 10 = worse pain possible)at 6 hours post-operatively

SECONDARY OUTCOMES:
Total post-operative opioid analgesic requirements | in the first 48 hours post-operatively or until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Saccardi, M.D., Ph.D., Principal Investigator — University of Padova; Massimo Micaglio, M.D., Principal Investigator — Azienda Ospedaliera Padova; Matteo Parotto, M.D., Ph.D., Principal Investigator — University of Padova
Locations (1):
- Azienda Ospedaliera-Università Padova, Padua, Padova, Italy